CLINICAL TRIAL: NCT06074757
Title: Open Label Sequential Dosing Single Ascending Dose of Four Cohort and Multiple Dose of One Cohort Pharmacokinetics Tolerability and Safety of Fulvestrant Injection as Test Product KSHN001034 vs Reference Product FASLODEX®
Brief Title: Open Label, Sequential Dosing , Single Ascending Dose and Multiple Dose Safety Tolerability and Pharmacokinetic Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kashiv BioSciences, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KSHN001034
Record Dates: First submitted 2023-08-21; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Intervention Model Description: open label, sequential dosing , single ascending dose and multiple dose pharmacokinetic , safety , tolerability study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- cohort 1 (Other): Test (25mg) vs RLD (500mg) to assess the safety and tolerability of the test dose
  Interventions: Drug: Fulvestrant injection
- cohort 2 (Experimental): Test 100 mg
  Interventions: Drug: Fulvestrant injection
- cohort 3 (Experimental): Test 250 mg
  Interventions: Drug: Fulvestrant injection
- cohort 4 (Experimental): Test 500mg
  Interventions: Drug: Fulvestrant injection

INTERVENTIONS:
Drug: Fulvestrant injection — phosphate ester of fulvestrant for test arm
  Other Names: faslodex

SUMMARY:
The goal of this clinical trial is to learn the comparative pharmacokinetic parameters between the test product and the Reference listed drug in healthy female volunteers

The main question[s] it aims to answer are:

* To assess the sequential dose exposure safety and tolerability of KSHN001034 injection in healthy female subjects after single ascending doses from 25 mg to 500 mg and multiple doses of maximum tolerable dose from single ascending dose
* To assess dose showing comparative bioavailability of KSHN001034 injection in comparison with Faslodex®.

DETAILED DESCRIPTION:
Single ascending dose (SAD) of four cohorts (01, 02, 03, and 04) for the test product (25, 100, 250, and 500 mg, respectively).

Subjects who will participate in cohort no. 01 (N= 18 subjects) will be randomized to receive a single dose of the test product 25 mg (N= 10 subjects) or a single dose of the reference product 500 mg (N= 08 subjects). The randomization ratio will be 5:4 for T: R Study Part II: Multiple doses of three treatment arms will be administered in one cohort (N= 32, parallel design).

• Two treatment arms of the test product: T1: the dose lower than maximum tolerated dose (MTD-1) determined in Study Part I, N=12 subjects.

T2: maximum tolerated dose determined in Study Part I, N=12 subjects.

• One treatment arm of the reference product: R: 500 mg, N= 08 subjects The randomization ratio will be 3:3:2 for T1:T2: R]

ELIGIBILITY:
Inclusion Criteria:

* The subject is healthy female adult of population aged between 40 to 60 years old (inclusive) at screening.
* The subject has a body weight not less than 50 Kg and according to the BMI range (18.5 - 30 Kg/m2)6 (inclusive) at screening.
* The subject is fully vaccinated for COVID-19 at least two weeks ago, as checked at screening.

  -. The subject is physically and mentally healthy as judged by means of medical and standard laboratory examinations at screening.
* The findings of the subject are within the range of clinical acceptability in medical history, and physical examination, and laboratory results "other than RBC indices (MCH, MCV and MCHC), and hemoglobin, " within "normal ranges" for the laboratory tests performed or abnormalities considered insignificant and justified by the principal/clinical sub- investigator at screening.
* The subject results are within normal range or ± 5% of medical lab reference range for all RBC indices (MCH, MCV and MCHC) and hemoglobin, at screening

  -. The subject's platelets count is within medical lab reference range at screening.
* The subject has a normal ECG (12 leads), including normal QTc (below 440 msec), at screening

  * The subject's chest X-ray, performed within 6 months before screening (if available) or at screening, is normal or considered clinically acceptable with no evidence of ongoing or past serious infections, as per the investigator judgment at screening.
  * The subject vital signs in sitting position are within the following ranges at screening, and on admission day (before admission):

Blood Pressure:

Systolic: (90 - 140) mmHg Diastolic: (60-90) mmHg Body Temperature: (36.1 - 37.2) ºC Pulse rate: 60 to 100 beat per minute. Respiratory rate: 12-18 bpm.

* Kidney function tests (Creatinine, Potassium and Sodium) are within the medical lab reference range and kidney function tests (Blood Urea Nitrogen, and uric acid) are considered clinically acceptable as per the investigator judgment at screening. If creatinine is below the lower normal limit while the other parameters are normal, it will be considered as clinically not significant unless otherwise judged by the investigator.
* Liver function tests (AST, ALT, GGT, and bilirubin (total, direct, and indirect)) results are within the medical lab reference ranges and liver function tests (Alkaline phosphatase, total protein, and albumin) are considered clinically acceptable as per PI / SI judgment at screening.

Exclusion Criteria:

* The subject has an evidence of psychiatric disorder, antagonistic personality, poor motivation, emotional or intellectual problems likely to limit the validity of the consent to participation in the study or limit the ability to comply with the protocol requirements, as determined by the principal investigator/clinical Sub-investigator at screening or on admission day (before admission).
* The subject has a known history or presence of any clinically significant abnormality / pathology / disease in any of the body systems, as checked at screening or on admission day (before admission).
* The subject has a clinically significant history or presence of any clinically significant gastrointestinal pathology (e.g. chronic diarrhea, active inflammatory bowel disease), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting), short bowel syndrome, upper gastrointestinal surgery including gastric resection, or other conditions known to interfere with the metabolism or excretion of the drug as determined by the principal investigator/clinical sub-investigator at screening or on admission day (before admission).
* The subject has a history of allergy or major allergic reactions or known allergy/ hypersensitivity to the drug under investigation (Fulvestrant), or to any of the excipients (ethanol, benzyl alcohol, benzyl benzoate, castor oil refined), as checked at screening
* The subject has a history of hypersensitivity to heparin as checked at screening.
* The subject has a history of vaginal bleeding or discharge, bleeding diatheses, thrombocytopenia or taking anticoagulant treatment as checked at screening.
* The subject has symptoms suggestive of COVID-19 as judged by the principal investigator/clinical sub-investigator at screening or admission day (before admission).

The subject is pregnant or nursing (lactating) women, where pregnancy is defined as the state of the female after conception and until the termination of gestation, confirmed by a positive serum pregnancy test at screening or on admission day (before admission).

* The subject has consumed or does not agree to abstain from consuming any beverages or food containing alcohol from screening until donating the last PK sample of the study cohort, as checked at screening or on admission day (before admission).
* The subject does not agree to abstain from consuming any beverages or food containing methylxanthines e.g. caffeine (coffee, tea, cola, energy drinks, chocolate, …etc) for at least 24 hours prior to each dosing and for 24 hrs after each dosing, as checked at screening or on admission day (before admission).
* The subject has taken any prescribed drugs within four weeks preceding first study drug administration or doesn't agree on not taking them until donating last PK sample of the study cohort, as checked at screening or on admission day (before admission).

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — healthy female
Enrollment: 48 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-09-10 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
safety and tolerability | 0-4 days
  To assess the dose exposure safety and tolerability of KSHN001034 injection in healthy female subjects after single ascending doses from 25 mg to 500 mg in sequential dosing and multiple doses of maximum tolerable dose from single ascending dose in parallel dosing
bioavailability | 0-28 days
  To assess dose showing comparative bioavailability of KSHN001034 injection in comparison with Faslodex®.

SECONDARY OUTCOMES:
fluctuation index and pharmacokinetics | 0-28 days
  To assess fluctuation index of Test vs RLD in multiple doses and To assess comparative pharmacokinetics of KSHN001034 injection in comparison with Faslodex

CONTACTS AND LOCATIONS:
Overall Officials: Dr Uday Harle, Phd medicine, Study Director — Kashiv biosciences
Locations (1):
- Triumpharma Cro, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No